| Evaluation of a peer-led web | -based intervention | for safe usage of d | lating |
|---|---|---|---|
| applications in Hong | Kong: a randomize | d controlled trial | |

## **Statistical Analysis Plan**

August 2018

(Version 1. Dated 17.08.2018)

Principle Investigator: Dr. William Wong
Address: Department of Family Medicine and Primary Care, 161 Ap Lei Chau Main
Street, Ap Lei Chau, Hong Kong
Co-Investigators: Tsz Hei Stephanie Lau, Dr. Julie Chen

## Statistical Methods

The demographics were described and differences in baseline were assessed using chi-square tests for categorical variables for e.g. age, gender and sexual orientation; and, *t*-test for scaled outcomes. The satisfaction of the intervention at post-intervention was analysed using chi-square test. ITT with the "last observation carried forward" values was adopted. Due to the skewness distribution of the outcomes, the differences of intervention at follow-ups were assessed using Mann-Whitney U-test. Univariate linear regression and multiple linear model was used to evaluate the significant factors between the intervention and control groups and after the adjustment of baseline outcome measurements respectively. All data were entered, cleaned and analysed using SPSS (Version 25) and significant tests were set at P-values <0.05.